CLINICAL TRIAL: NCT04563299
Title: Effect on Pain and Inflammation With DEXTENZA Treatment in Patients Undergoing Intravitreal Anti-VEGF Injections
Acronym: DETeR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subject Enrollment
Sponsor: Retina Vitreous Associates of Florida (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, David Eichenbaum, Principal Investigator, Retina Vitreous Associates of Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DETeR
Record Dates: First submitted 2020-09-10; First posted 2020-09-24 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: This is an investigator initiated prospective open-label, within-patient, masked, randomized study in patients with neovascular AMD, DME, or RVO undergoing bilateral anti-VEGF injections. Within the respective cohorts, one eye per patient will be randomized to receive either an intracanalicular dexamethasone insert or the control treatment at each injection visit.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the survey administrator are masked to the treatment assignment in each eye.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza (Experimental): Dextenza (Dexamethasone Ophthalmic Insert 0.4 mg)
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Topical Corticosteroids (Active Comparator): Topical corticosteroids (prednisolone acetate 1%) QID tapered over 4 weeks (QID/ 1 week, TID/ 1 week, BID/1 week, QD/ 1 week).
  Interventions: Drug: Prednisolone Acetate

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — All eyes (n=40) will receive anti-VEGF injections for the treatment of AMD, DME and macular edema secondary to RVO. Twenty eyes (one eye per patient) will be randomized to receive Dextenza. The contra-lateral eye (Control) will receive a sham dilation.
  Arms: Dextenza
Drug: Prednisolone Acetate — All eyes (n=40) will receive anti-VEGF injections for the treatment of AMD, DME and macular edema secondary to RVO. Twenty eyes (one eye per patient) will be randomized to receive Dextenza. The contra-lateral eye (Control) will receive topical corticosteroids (prednisolone acetate 1%) QID tapered over 4 weeks (QID/ 1 week, TID/ 1 week, BID/1 week, QD/ 1 week).
  Arms: Topical Corticosteroids

SUMMARY:
This is an investigator initiated prospective open-label, within-patient, masked, randomized study in patients with neovascular AMD, DME, or RVO undergoing bilateral anti-VEGF injections. Patients will be randomized into two cohorts (Cohort 1 and Cohort 2) and then followed for 3 consecutive injection visits. Treatment will be rendered at each injection visit based on the individualized routine established anti-VEGF injection interval for each patient.

DETAILED DESCRIPTION:
This is an investigator initiated prospective open-label, within-patient, masked, randomized study in patients with neovascular AMD, DME, or RVO undergoing bilateral anti-VEGF injections. Patients will be randomized into two cohorts (Cohort 1 and Cohort 2) and then followed for 3 consecutive injection visits. Treatment will be rendered at each injection visit based on the individualized routine established anti-VEGF injection interval for each patient.

Within the respective cohorts, one eye per patient will be randomized to receive either an intracanalicular dexamethasone insert or the control treatment at each injection visit. Cohorts are as follows:

Cohort 1:

Total N= 40 eyes (20 patients). Twenty eyes (one eye per patient) will be randomized to receive an intracanalicular dexamethasone insert. The contra-lateral eye (Control) will receive a sham dilation.

Cohort 2:

Total N= 40 eyes (20 patients). Twenty eyes (one eye per patient) will be randomized to receive an intracanalicular dexamethasone insert. The contra-lateral eye (Control) will receive topical corticosteroids (prednisolone acetate 1%) QID tapered over 4 weeks (QID/ 1 week, TID/ 1 week, BID/1 week, QD/ 1 week).

In eyes randomized to either DEXTENZA or sham dilation, DEXTENZA insertion or sham dilation will be performed prior to injection.

In eyes randomized to either DEXTNEZA or topical steroids, eyes randomized to DEXTENZA will receive insertion prior to injection. Eyes randomized to topical steroid therapy (Control) will receive 1 drop of prednisolone acetate 1% pre-injection and the remaining 3 drops of prednisolone acetate 1% post injection. Control eyes will follow tapered dosing over 4 weeks (QID/ 1 week, TID/ 1 week, BID/1 week, QD/ 1 week) to ensure dose matching between DEXTENZA and Control in Cohort 1.

Pain will be rated at 6 time points: (1) prior to any treatment, (2) after anesthesia, (3) after intravitreal injection, (4) 6 hours by telephone (+/- 2 hours), (5) 24 hours by telephone (+/-3 hours) and (6) 3-6 days at assessment visit. Pain will be evaluated by survey administrators masked to treatment assignment. Patient comfort (right eye vs left eye) will be assessed at each patient visit by masked survey administrator. Anterior cell count and anterior cell flare assessment will be conducted at 3-6 days following each intravitreal injection visit. There will be a final patient preference survey performed.

ELIGIBILITY:
Inclusion Criteria: A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* Patients diagnosed with neovascular AMD, DME or macular edema secondary to RVO undergoing anti-VEGF injections in both eyes.
* > 18 years old
* Able to provide signed written consent prior to participation in any study-related procedures.

Exclusion Criteria: A patient who meets any of the following criteria will be excluded from the study:

* Prescription and OTC ophthalmic mast cell stabilizers and antihistamines within 21 days prior to Screening and throughout the study period (systemic mast cell stabilizers are allowed, and systemic antihistamines are permitted)
* Use of any topical prescription ophthalmic medications (including cyclosporine [Restasis®, Cequa®] or topical lifitegrast [Xiidra®], steroids, nonsteroidal anti- inflammatory drugs [NSAIDs]within 7 days or during study period
* Participation in any drug or device clinical investigation within 30 days prior to study entry and/or during the study period.
* Anterior chamber cells present at time of enrollment
* History of cauterization of the punctum
* Any punctum inflammation or dacryocystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Mean Change in Pain Scores | As assessed at Baseline Visit, 6 hours (+/- 2 hours), 24 hours (+/- 3 hours), and at 3-6 days after Injection Visit 1, Injection Visit 2, and Injection Visit 3
  As measured by a 10-point standardized pain scale (1 = no pain, 10 = worst pain)

SECONDARY OUTCOMES:
Overall Proportion of Eyes with Absence of AC Cell/Flare (Score of 0) | Assessed 3-6 days following Injection Visit 1, Injection Visit 2, and Injection Visit 3
  As measured using SUN criteria
Proportion of eyes with absence of AC cells/flare (score of 0) | Assessed at 3-6 days following Injection Visit 1, Injection Visit 2, and Injection Visit 3 by anti-VEGF type (ranibizumab, aflibercept, brolucizumab, or bevacizumab)
  As measured using SUN criteria
Correlation of pain scale outcomes with absence or presence of AC cell count and flare scores | Assessed at 3-6 days after Injection Visit 1, Injection Visit 2, and Injection Visit 3
  As measured using pain scale outcomes with absence or presence of AC cell count and flare scores
Mean Change in pain scores | As assessed at Baseline Visit, 6 hours (+/- 2 hours), 24 hours (+/- 3 hours), and at 3-6 days after Injection Visit 1, Injection Visit 2, and Injection Visit 3
  As measured by a 10-point standardized pain scale (1 = no pain, 10 = worst pain)
Patient Comfort | As assessed at Baseline Visit, 6 hours (+/- 2 hours), 24 hours (+/- 3 hours), and at 3-6 days after Injection Visit 1, Injection Visit 2, and Injection Visit 3
  As measured by masked survey administrator
Mean Change in Tear Break-up Time | As assessed at Baseline Visit, Injection Visit 1, Injection Visit 2, Injection Visit 3, and the Final Post-Injection Follow-up Visit (up to 24 weeks)
  As measured by the tear break-up time
Mean Change in Snellen and Pinhole Acuity | As assessed at Baseline Visit, Injection Visit 1, Injection Visit 2, and Injection Visit 3, and the Final Post-Injection Follow-up Visit (up to 24 weeks)
  As measured by the ETDRS visual acuity chart
Mean change in IOP | As assessed at Baseline Visit, Injection Visit 1, Injection Visit 2, and Injection Visit 3, and the Final Post-Injection Follow-up Visit (up to 24 weeks)
  As measured by using a Tono-pen
Patient Preference | As assessed at the Final Post-Injection Follow-up Visit (up to 24 weeks)
  As measured by modified COMTOL
Incidence and severity of adverse events | As assessed at Baseline, 6 hours (+/- 2 hours), 24 hours (+/- 3 hours), 3-6 days after Injection Visit 1, Injection Visit 2, and Injection Visit 3, and the Final Post-Injection Follow-up Visit (up to 24 weeks)
  As measured by the incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: David Eichenbaum, MD, Principal Investigator — Retina Vitreous Associates of Florida
Locations (1):
- Retina Vitreous Associates of Florida, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No